CLINICAL TRIAL: NCT04536129
Title: Effects of Topical Low Dose Preservative-free Hydrocortisone on Intraocular Pressure in Patients With and Without Glaucoma
Brief Title: Effects of Topical Low Dose Preservative-free Hydrocortisone on Intraocular Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Molise (Other)
Collaborators: Medivis SRL (Industry)
Responsible Party: Principal Investigator, Ciro Costagliola, Full Professor in Ophthalmology, University of Molise
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTS 11/2019
Record Dates: First submitted 2020-08-27; First posted 2020-09-02 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Ocular Surface Disease; Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: glaucoma (Experimental): OSD patients with glaucoma
  Interventions: Drug: Hydrocortisone (CORTIVIS ®)
- Group B: no glaucoma (Active Comparator): OSD patients without glaucoma
  Interventions: Drug: Hydrocortisone (CORTIVIS ®)

INTERVENTIONS:
Drug: Hydrocortisone (CORTIVIS ®) — Once enrolled all the patients had to instill topical low dose (1,005 mg) preservative-free hydrocortisone (CORTIVIS ®- Medivis, Catania, Italy) 2 times daily in each eye for two weeks.

SUMMARY:
Evaluation of the safety and efficacy of hydrocortisone eye drops in the treatment of OSD (ocular surface disease) patients with and without glaucoma.

DETAILED DESCRIPTION:
The ocular surface comprises the cornea, conjunctiva, eyelids and lacrimal glands and any disorder in these structures can be classified as an ocular surface disorder (OSD). OSD includes Dry Eye Disease (DED), blepharitis and meibomian gland dysfunction (MDG), allergic eye diseases (AED), chemical and thermal burns; all these conditions can severely affect eyesight and quality of life, and sometime even blindness. Patients with OSD can develop photophobia, corneal scarring, intermittent blurred vision, pain, limited ability to perform daily activities, reduced vitality, poor general health and, in many cases, depression.

Glaucoma, one of the leading causes of irreversible blindness, is an optic neuropathy characterized by thinning of retinal nerve fiber layer and increase of optic disc cupping , whose main risk factor is closely related to the intraocular pressure (IOP) levels. Thus, the management of the disease consists in the lowering IOP through medical, laser or surgical therapy . However, IOP reduction is most commonly achieved using topical ocular medications, which often contain preservatives employed to maintain stability and sterility of the product. Preservatives can be associated with undesirable adverse effects such as allergy, local irritation and inflammation . The long-term use of anti-glaucoma medications produces several alterations of ocular surface components, especially at the conjunctival level where epithelial modifications, dendritic cell activation, conjunctiva-associated lymphoid tissue activation, and goblet cell (GCs) loss easily occur GCs play crucial tasks in the homeostasis of the ocular surface being the main source of mucoproteins, essential to maintain tear film stability. Thus, the loss of GCs progressively leads to the happening of an iatrogenic OSD . Moreover, advancing age is a significant risk factor for both OSD and glaucoma, further complicated by treatments for each condition, which can interact among them and yield counterproductive effects . For these reason glaucoma is often associated with OSD .Ocular surface inflammation is crucial in the pathophysiology of OSD, therefore anti-inflammatory therapy, including corticosteroids, may be of benefit to OSD patients . However, in susceptible individuals steroid-induced glaucoma or ocular hypertension can occur after steroid use. Individuals who develop an increase in IOP following steroid use are referred to as "steroid responders" . In a recent study Kallab et al. have found that dry eye treatment with low hydrocortisone dose reduced ocular inﬂammation without inducing increases in IOP ; glaucomatous patients were excluded from this study. Herein we evaluate the safety and efficacy of hydrocortisone eye drops in the treatment of OSD patients with and without glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* age of at least 18 years
* diagnosis of OSD (Ocular Surface Disease)
* normal ophthalmic ﬁndings except history of OSD for at least 3 months, and current therapy with topical lubricants for at least 3 months
* POAG (primary open-angle glaucoma ) patients on medical therapy

Exclusion Criteria:

* clinically signiﬁcant slit lamp ﬁndings at screening visit except OSD
* participation in a clinical trial in the 4 weeks preceding the screening visit
* symptoms of a clinically relevant illness in the 3 weeks before the screening visit
* presence/ history of a severe medical or surgical condition
* intake of parasympathomimetic or antipsychotic drugs
* wearing of contact lenses
* previous refractive laser surgery (e.g photorefractive keratectomy-PRK, laser assisted in situ keratomileusis-LASIK, etc.)
* history of IOP increase caused by systemic or topical treatment with corticosteroids
* IOP greater than 22 mmHg
* treatment with corticosteroids in the 4 weeks preceding the study
* types of glaucoma other than POAG
* ocular infection or clinically signiﬁcant inﬂammation
* ocular surgery in the 3 months preceding the study
* Sjögren's syndrome, Stevens-Johnson syndrome
* history of allergic conjunctivitis
* pregnancy, planned pregnancy or lactating
* known hypersensitivity to any component of study medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure(IOP) | 2 weeks
  IOP evaluation at time zero (T0), after 1 (T1) and two weeks of therapy (T2).
OSDI (Ocular Surface Disease Index) questionnaire | 2 weeks
  OSDI record at time zero (T0), after 1 (T1) and two weeks of therapy (T2).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Molise, Campobasso, Italy

REFERENCES:
- [Result] Khanna RC. Ocular surface disorders. Community Eye Health. 2017;30(99):S1-S2. No abstract available. PMID 29849435
- [Result] Craig JP, Nelson JD, Azar DT, Belmonte C, Bron AJ, Chauhan SK, de Paiva CS, Gomes JAP, Hammitt KM, Jones L, Nichols JJ, Nichols KK, Novack GD, Stapleton FJ, Willcox MDP, Wolffsohn JS, Sullivan DA. TFOS DEWS II Report Executive Summary. Ocul Surf. 2017 Oct;15(4):802-812. doi: 10.1016/j.jtos.2017.08.003. Epub 2017 Aug 8. PMID 28797892
- [Result] Lanza M, Gironi Carnevale UA, Mele L, Bifani Sconocchia M, Bartollino S, Costagliola C. Morphological and Functional Evaluation of Oral Citicoline Therapy in Chronic Open-Angle Glaucoma Patients: A Pilot Study With a 2-Year Follow-Up. Front Pharmacol. 2019 Sep 26;10:1117. doi: 10.3389/fphar.2019.01117. eCollection 2019. PMID 31611797
- [Result] Mohammed I, Kulkarni B, Faraj LA, Abbas A, Dua HS, King AJ. Profiling ocular surface responses to preserved and non-preserved topical glaucoma medications: A 2-year randomized evaluation study. Clin Exp Ophthalmol. 2020 Sep;48(7):973-982. doi: 10.1111/ceo.13814. Epub 2020 Jul 27. PMID 32564453
- [Result] Rossi GC, Pasinetti GM, Scudeller L, Bianchi PE. Ocular surface disease and glaucoma: how to evaluate impact on quality of life. J Ocul Pharmacol Ther. 2013 May;29(4):390-4. doi: 10.1089/jop.2011.0159. Epub 2012 Dec 7. PMID 23215770
- [Result] Rossi GC, Pasinetti GM, Scudeller L, Raimondi M, Lanteri S, Bianchi PE. Risk factors to develop ocular surface disease in treated glaucoma or ocular hypertension patients. Eur J Ophthalmol. 2013 May-Jun;23(3):296-302. doi: 10.5301/ejo.5000220. Epub 2012 Dec 17. PMID 23335308
- [Result] Kallab M, Szegedi S, Hommer N, Stegmann H, Kaya S, Werkmeister RM, Schmidl D, Schmetterer L, Garhofer G. Correction to: Topical Low Dose Preservative-Free Hydrocortisone Reduces Signs and Symptoms in Patients with Chronic Dry Eye: A Randomized Clinical Trial. Adv Ther. 2020 Jan;37(1):342-343. doi: 10.1007/s12325-019-01190-3. PMID 31823206
- [Derived] Filippelli M, dell'Omo R, Gelso A, Rinaldi M, Bartollino S, Napolitano P, Russo A, Campagna G, Costagliola C. Effects of topical low-dose preservative-free hydrocortisone on intraocular pressure in patients affected by ocular surface disease with and without glaucoma. Graefes Arch Clin Exp Ophthalmol. 2022 Jan;260(1):247-253. doi: 10.1007/s00417-021-05345-3. Epub 2021 Aug 18. PMID 34406502